CLINICAL TRIAL: NCT02749617
Title: A Pilot Study Investigating Apixaban and Dexamethasone InterAction in Multiple Myeloma
Acronym: ADAM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was stopped due to lack of enrollment.
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Agnes Lee, Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H14-01652
Record Dates: First submitted 2016-03-30; First posted 2016-04-25 (Estimated); Results first posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-07

CONDITIONS: Anti-Xa Activity
MeSH Terms: interventions — apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- apixaban (Experimental): apixaban 2.5 mg PO BID
  Interventions: Drug: apixaban

INTERVENTIONS:
Drug: apixaban — 2.5 mg PO BID
  Other Names: Eliquis

SUMMARY:
This pilot study will investigate the impact of dexamethasone (DEX) on anti-Xa levels in participants taking apixaban 2.5 mg twice a day by mouth (PO BID). Investigators propose a prospective, cohort study of 24 participants with multiple myeloma, in whom a lenalidomide-dexamethasone (LEN-DEX)-based myeloma treatment regimen is indicated. Eligible participants will initiate thromboprophylaxis with apixaban prior to starting their DEX-containing regimen and continue until the end of cycle 3. Anti-Xa levels, D-Dimer and plasma drug concentration will be measured.

This pilot study looks to investigate this potential interaction between apixaban and dexamethasone to see if it warrants further investigation in a larger study.

The sample size of 24 provides 90% power to detect a primary outcome of ≥ 50% reduction in peak anti-Xa levels from baseline. Secondary outcomes include changes in plasma apixaban levels, D-dimer, and symptomatic venous thromboembolism (VTE) and bleeding during a 3-month treatment period.

DETAILED DESCRIPTION:
Study has terminated due to poor enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of multiple myeloma according to criteria of the International Myeloma Working Group
* Patients in whom a LEN-DEX-based treatment regimen is indicated
* Adult patients ≥ 19 years of age who are able to freely provide informed consent

Exclusion Criteria:

* Concomitant antiplatelet or anticoagulant use
* Calculated creatinine clearance < 30 mL/min by Cockcroft-Gault formula
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 times upper limit of normal (ULN)
* Total bilirubin > 2 x ULN
* Thrombocytopenia < 50 x 10 gigalitres (Gl)
* High bleeding risk or spontaneously prolonged prothrombin time or activated partial thromboplastin time > 1.5 x ULN
* Body weight <50 or >120 kg
* Concomitant use of CYP3A4 or p-glycoprotein inducers or inhibitors
* Use of Ginkgo biloba or St. John's Wort within 14 days before first dose of study drug
* Dexamethasone use within last 3 months
* Women of Childbearing potential without proper contraceptive measures, pregnancy or breast feeding
* Life expectancy less than 3 months
* Inability to swallow or issues with malabsorption
* Any other medical, social, logistical, geographical or psychological factors, which in the opinion of the investigator, would prohibit follow-up, compliance and study completion

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-08-09 (Actual); Primary Completion 2018-01-03 (Actual); Study Completion 2019-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Agnes YY Lee, MD MSc FRCPC, Principal Investigator — University of British Columbia, Division of Hematology
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Apixaban
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Apixaban
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 2

OUTCOME MEASURES:

1. Primary Outcome: Anti Xa Activity
Description: serial anti Xa activity
Time Frame: 3 months
Population: Lack of data.
Arm/Group | Apixaban
Number analyzed (Participants) | 0

2. Secondary Outcome: Plasma Apixaban Levels
Description: Due to lack of enrollment, plasma apixaban levels were not analyzed
Time Frame: 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Apixaban
All-Cause Mortality (participants affected / at risk) | 2/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apixaban (N=2)
Nose Bleed (Blood and lymphatic system disorders) | 1 (3)
Nausea (General disorders) | 1 (1)
Flu-like Symptoms (General disorders) | 1 (1)
Diarrhea (General disorders) | 1 (1)
Pseudomonas aerugionosa (General disorders) | 1 (1)
Skin Itchiness (General disorders) | 1 (3)
Low Energy (General disorders) | 1 (1)
Back right-sided buttock pain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/17/NCT02749617/Prot_SAP_000.pdf